CLINICAL TRIAL: NCT06989294
Title: Effect of Lean Leadership Training Program on Head Nurses' Lean Performance and Staff Nurses' Workplace Safety at Mansoura Children Hospital
Acronym: leadership
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Lean Leadership
Record Dates: First submitted 2025-05-07; First posted 2025-05-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-04

CONDITIONS: Safety Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lean Leadership and Staff Nurses' Workplace Safety (Experimental): Lean leadership is a modern concept for process optimization throughout the value chain that is focusing on making inefficiencies (waste) transparent and on altering these into value-adding activities, improve physical work environments for healthcare professionals and workplace safety. Workplace Safety is positive and healthy work environments as places where nurses are encouraged to be high performers, where resources are adequately used, and employees can achieve an organizational goal while staying safe.
  Interventions: Other: Lean Leadership

INTERVENTIONS:
Other: Lean Leadership — Lean leadership was doing the right things to increase revenues, satisfying customers and reducing costs by eliminating all activities that do not add value to the product or service. It has five dimensions, namely: continuous improvement, self-development, qualification development, Gemba walk and Hoshin Kanri.

SUMMARY:
Effect of Lean Leadership Training Program on Head Nurses' Lean Performance and Staff Nurses' Workplace Safety at Mansoura Children Hospital

DETAILED DESCRIPTION:
Many global healthcare challenges, such as infections, preventable errors, growing healthcare costs, and changing patient expectations, have a negative impact on health outcomes. Lean management provides a solution to these problems by reducing costs and eliminating waste . So, implementation of lean practices improves staff performance, adapt to new competitors, and foster flexibility. They are beneficial for economic growth. Research shows that lean practices improve knowledge and skills of head nurses, improve environmental quality, and create a safer and more productive work environment . This study will provide more focus on the value of lean leadership as a new approach to be implemented in Egyptian hospitals to improve leader's competencies, capacity, and skills in determining wastes in care processes by using lean tools and for continuous improvement. Also, it will help in enhancing workplace safety and to provide safe and appropriate care for patient which result in improving health care system as a general. Hence the present study aims to evaluate the effect of a lean leadership training program on workplace safety.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study.
* Head nurses have at least one year of job experience.

Exclusion Criteria:

* Agree to involve in the study. - Staff nurses have at least one year of job experience in the current job

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Staff Nurses' perception about work environment safety as assessed by Practice Environment Scale of the Nursing Work Index (PES - NWI | from start to finish, up to three month
  The Practice Environment Scale of the Nursing Work Index (PES-NWI) is an instrument, which measures the nursing practice environment - defined as factors that enhance or attenuate a nurse's ability to practice nursing skillfully and deliver high quality care.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Mansoura University, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alshyyab, M. A., FitzGerald, G., Ababneh, E. Y., Zghool, A. W., & Albsoul, R. A. (2023). Nurses' perceptions regarding the impact of teamwork on patient safety culture in the operating room: A qualitative study. Perioperative Care and Operating Room Management, 33, 100345.
- See also: Al-hadrawi R and Al-Abedi M. (2020). The impact of lean leadership on the creative work behavior: perceived organizational support as the moderator variable. An analytical study in the Iraqi health sector. International Journal of Psychosocial — https://www.researchgate.net/publication/347902923_Lean_Leadership